CLINICAL TRIAL: NCT06863389
Title: Comparison of Chen's U-suture Technique with Duct-to-Mucosa Anastomosis and Invagination Pancreaticojejunostomy After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: Chen'sUsuture1
Record Dates: First submitted 2025-02-24; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Chen's group: performing pancreaticojejunostomy by using Chen's U-suture technique
  Interventions: Procedure: Chen's U-suture technique
- Invagination group: performing pancreaticojejunostomy by using invagination method
  Interventions: Procedure: invagination
- Duct-to-Mucosa group: performing pancreaticojejunostomy by using duct-to-mucosa method
  Interventions: Procedure: Duct-to-Mucosa

INTERVENTIONS:
Procedure: Chen's U-suture technique — Initially, an approximately 2 cm cut edge of the pancreas remnant was mobilized and a incision of the jejunal loop was conducted slightly shorter than the pancreatic remnant. Using dual-needle 3-0 prolene suture for anastomosis, needle A went through the entire intestinal wall from the posterior wall about 1.5 cm away from the resection margin of the jejunum loop, then went through the superior boarder of the pancreas from posterior to anterior. To suture the anterior wall of the jejunum loop, the stitch next entered from the resection margin of the jejunum loop and kept it within the seromuscular layer from proximal to distal, and got out from about 1.5 cm away from the resection margin. Needle B repeated the aforementioned procedures with a parallel distance about 1.0 cm between needle A. Generally, the whole anastomosis needed two to four identical stitches. The stitches should overlap each other to reduce pancreatic leakage. Once all the stitches were finished and tighte
  Groups: Chen's group
Procedure: invagination — Firstly, using 3-0 silk sutures, the pancreatic capsule and the serosa of the jejunal loop were anastomosed interruptedly to constitute the posterior outer layer of the anastomosis. Secondly, a jejunotomy with an appropriate size was performed and the inner layer (including posterior and anterior) of invagination was formed by two 5-0 prolene sutures with a continuous running between the pancreatic parenchyma and the full-thickness jejunum. Thirdly, the anterior outer layer was sutured in line with the first step.
  Groups: Invagination group
Procedure: Duct-to-Mucosa — Briefly, Duct-to-Mucosa should make a opening matched to the pancreatic duct and was also performed by two layers. One was the outer layer in both the anterior and posterior walls of the anastomosis which were formed by interrupted 3-0 silk sutures betweent the pancreatic capsule and the jejunal serosa. The other was the inner layer performed in eight to twelve stitches from pancreatic duct to jejunal mucosa with 5-0 prolene sutures.
  Groups: Duct-to-Mucosa group

SUMMARY:
Data of patients treated with pancreaticoduodenectomy in 21 hospitals from January 2014 to December 2019 were retrospectively collected and classified to Chen's group, duct-to-mucosa group and invagination group according to different pancreaticojejunostomy. Propensity score matching analysis was performed to balance the baseline differences among three groups. The surgical outcomes were compared. Independent risk factors for postoperative pancreatic fistula were confirmed by logistic regression analysis, and subgroup analysis was also conducted.

ELIGIBILITY:
Inclusion Criteria:

* open pancreaticoduodenectomy
* Chen's U-suture technique or invagination or duct-to-mucosa anastomosis

Exclusion Criteria:

* missing data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent open pancreaticoduodenectomy during the period from January 1, 2014 to December 31, 2019 at 21 hospitals in China were restrospectively recruited. All patients underwent standard open pancreaticoduodenectomy with Child reconstruction which were performed by senior hepato-pancreato-biliary surgeons who performed over 200 pancreaticoduodenectomy per year. According to different PJ, patients were divided into three groups: Chen's, IG, DTM.
Sampling Method: Non-Probability Sample
Enrollment: 5788 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
postoperative pancreatic fistula | postoperative 30 days
  Postoperative pancreatic fistula was diagnosed and graded in accordance with the 2016 update definition of the International study group (ISGPS)